CLINICAL TRIAL: NCT06971900
Title: A Phase 2a, Blinded, Randomized, Placebo-Controlled Study of PORT-77 Administered Orally to Adults With Erythropoietic Protoporphyria
Brief Title: GATEWAY: A Phase 2a Study of PORT-77 in Adults With Erythropoietic Protoporphyria
Acronym: EPP
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Portal Therapeutics, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PORT-77-201
Record Dates: First submitted 2025-04-03; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Erythropoietic Protoporphyria (EPP)
Keywords: PORT-77; EPP; erythropoietic protoporphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PORT-77 (Experimental): Active
  Interventions: Drug: PORT-77
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PORT-77 — Active oral dose form
  Arms: PORT-77
Drug: Placebo — Matching inactive oral dose form
  Arms: Placebo

SUMMARY:
A Phase 2a study of PORT-77 in adults with erythropoietic protoporphyria (EPP)

ELIGIBILITY:
Major Inclusion Criteria:

* BMI ≥18.0 and ≤35.0 kg/m2 and weight ≥50 kg
* Known diagnosis of EPP and is currently symptomatic even if receiving treatment for EPP, including afamelanotide.
* Willing and able to avoid exposure to sunlight when outside of the clinical research site.
* Willing and able to follow protocol-specified contraception guidance.
* Able to read and understand English
* Able to understand the study procedures as described in the ICF and is willing and able to comply with the study requirements.

Major Exclusion Criteria:

* Is mentally or legally incapacitated
* History or presence of any illness or clinically significant medical or psychiatric condition or disease that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
* History of gastrointestinal condition, including surgeries, which may affect absorption after oral administration.
* History of cancer, with the exception of cutaneous non-melanoma skin cancer (basal or squamous cell carcinoma).
* Participation in another clinical study within 28 days or within 5 half-lives (if known), prior to screening
* Unable to refrain from or anticipates the use of medications/supplements known to confound PORT-77 beginning 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study drug and throughout the study.
* Estimated glomerular filtration rate <80 mL/min/1.73 m2 using the CKD-EPI equation at screening
* Hepatic impairment, with alanine aminotransferase, aspartate aminotransferase, or total bilirubin >1.5 x ULN at screening
* Female participant with a positive pregnancy test at screening or who is breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Plasma PPIX level | 9 Days
  Change over the course of the study in plasma PPIX concentrations

SECONDARY OUTCOMES:
Evaluate safety and tolerability of 2 different dose regimens of PORT-77 | 9 Days
  Safety and tolerability over the course of the study, as assessed by adverse events (AEs) and laboratory results
Cmax | Predose and 1, 2, 3, 4, 6, 8, 12 hours post dose
  Maximum measured concentration of PORT-77 in plasma (Cmax).
Tmax | Predose and 1, 2, 3, 4, 6, 8, 12 hours post dose
  Time from dosing to maximum measured concentration of PORT-77 in plasma
AUC0-last | Predose and 1, 2, 3, 4, 6, 8, 12 hours post dose
  Area under the concentration-time curve of of PORT-77 in plasma over the time interval from 0 to the time of the last quantifiable data point.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Portal Therapeutics, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided